CLINICAL TRIAL: NCT03653377
Title: Survey on the Human Papilloma Virus Vaccination in Girls With Cystic Fibrosis Followed in Cystic Fibrosis (CF) Center in France
Brief Title: Human Papilloma Virus Vaccination in Girls With Cystic Fibrosis (VACCIN-HPV-MUC2)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0144; 2018-A01314-51 (Other: ID-RCB)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Mucoviscidosis
Keywords: mucoviscidosis; Human Papilloma Virus; Vaccination; Young girl
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with self-administered questionnaire
  Interventions: Other: Self administrated questionnaire

INTERVENTIONS:
Other: Self administrated questionnaire — Questionnaires are distributed to patients with their parents during their visit to the CF center.

SUMMARY:
Background The main risk factor for cervical cancer is the infection by human papillomavirus (HPV). Vaccination against HPV, offered to all girls aged 11 to 14 is an effective method of prevention against cervical pathology. Despite this, vaccination coverage against HPV remains low in France. A proportion of women with cystic fibrosis may be involved in transplantation, a factor associated with a higher risk of HPV carriage and cervical pathology. An over-risk of cervical pathology would also be present in women with non-transplanted cystic fibrosis. Particular attention to vaccination should therefore be included in this population.

Objectives of the study The main objective of the study is to estimate the frequency of HPV vaccination in young girls with CF over 9 years and followed in a pediatric CF center.

The secondary objectives are to know:

* The type of vaccine used (bivalent / quadrivalent / nonavalent)
* The proportion of vaccinated girls with respect of the vaccination schedule (number of injections / spacing between doses)
* Reasons for non-use of vaccination

Study design The study will last 12 months. It is a cross-sectional, non-interventional, multicenter conducted by self-administered questionnaire.

Population

* young girls aged 9 years or older with Cystic fibrosis
* Followed in a pediatric or mixed CF center in the France (Rhone-Alpes Auvergne Region and Ile de France Region)
* With parents who did not object to participation in the study

Number of subject: 62 patients

Expected results

* Knowledge of HPV vaccination coverage in young girls with CF.
* Sensitization of patients, their parents and health professionals to HPV vaccination. Understand the barriers and reasons for refusing vaccination to promote actions to improve immunization coverage.

ELIGIBILITY:
Inclusion Criteria:

* young girls aged 9 years or older
* patients with Cystic Fibrosis
* patients followed in a pediatric or mixed CF center in the France (Rhone-Alpes Auvergne Region and Ile de France Region)
* patients with parents who did not object to participation in the study

Exclusion Criteria:

-patients who refuse to answer to the self-administrated questionnaire

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort of minor girls with cystic fibrosis older than 9 years, followed in a pediatric Mucoviscidosis Resource and Competence Center (MRCC).
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
HPV vaccination | Baseline
  The outcome measure is having HPV vaccination. This information is collected through a self-questionnaire, completed by the patients or their parents, during a visit to the CF center

CONTACTS AND LOCATIONS:
Overall Officials: Christine ROUSSET-JABLONSKI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Service Mucoviscidose, Pneumologie, Bron
  - Hôpital d'Estaing, Clermont-Ferrand
  - Pôle Couple / Enfant, Grenoble
  - CRCM, Hôpital Robert Debré, Paris
  - CRCM, Hôpital Trousseau, Paris
  - CRCM, Institut Necker Enfants Malade, Paris
  - Centre de Ressources et de Compétences de la Mucoviscidose Adultes, Pierre-Bénite